CLINICAL TRIAL: NCT06910332
Title: The Effect of Shoulder Mobilization on Muscle Strength and Proprioception: a Randomized Double-blind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ACU-FTR-AOA
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy Male and Female Subjects
Keywords: mobilization; proprioception; strength; shoulder
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the shoulder mobilization group or the sham mobilization group, and they remain in their assigned group throughout the study. This design allows for a direct comparison of the acute effects of mobilization on muscle strength and proprioception.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization Group (Experimental): Participants receive passive shoulder joint mobilization targeting the glenohumeral joint.
  Interventions: Other: Joint mobilization
- Sham Group (Sham Comparator): Participants undergo a placebo procedure where the practitioner mimics the mobilization technique without applying actual joint movement or distraction.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Joint mobilization — Participants receive passive shoulder joint mobilization on the dominant-side glenohumeral joint. The mobilization includes inferior, anterior, and posterior glide techniques, each performed for 1 minute at a frequency of 0.5 Hz, with a 30-second rest between each mobilization. The participant is positioned comfortably to support the joint's range of motion.
  Other Names: Shoulder joint mobilization; Shoulder joint glides
  Arms: Mobilization Group
Other: Sham — In the sham intervention, the practitioner mimics the technique of shoulder mobilization but does not apply any actual movement or glide effect on the joint. The procedure is designed to closely resemble the real intervention in terms of duration, rhythm, and the practitioner's handling of the participant's shoulder. The practitioner will use superficial touch on the glenohumeral joint without applying any of the mobilizing forces necessary to move the joint.
  Other Names: Sham mobilization; Sham shoulder mobilization
  Arms: Sham Group

SUMMARY:
This randomized, double-blind study examines the acute effects of shoulder mobilization on muscle strength and proprioception in healthy individuals. Forty-eight participants (aged 18-25) were randomly assigned to either a mobilization or sham intervention group. Muscle strength and proprioception were assessed before and after treatment. The mobilization group received passive shoulder joint glides, while the sham group underwent a placebo procedure. The study aims to determine whether mobilization affects strength and proprioception immediately.

DETAILED DESCRIPTION:
Summary of the Study

This randomized, double-blind study investigates the acute effects of shoulder joint mobilization on muscle strength and proprioception in healthy individuals compared to a sham intervention.

Background:

The shoulder joint is highly mobile and prone to injury, with rehabilitation often including manual therapy techniques like joint mobilization. Mobilization may enhance joint stability, neuromuscular control, and proprioception by stimulating mechanoreceptors. However, its immediate effects on shoulder proprioception and strength remain unclear.

Methods:

Participants: 48 healthy university students (aged 18-25) randomly assigned to either the mobilization or sham group.

Assessments: Muscle strength (using a handheld dynamometer) and proprioception (laser pointer-assisted joint position reproduction test) were measured before and after the intervention.

Intervention: The mobilization group received passive shoulder joint glides, while the sham group underwent a placebo procedure without actual joint movement.

Conclusion:

This study aims to determine whether shoulder mobilization has immediate effects on proprioception and strength.

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students aged 18-25 years.

Exclusion Criteria:

* Individuals with orthopedic problems in the shoulder complex.
* Those who have undergone previous shoulder surgery.
* Participants with prior knowledge of joint mobilization techniques that could affect the sham intervention.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University Kerem Aydınlar Campus, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographic Data:
  Age and gender,
  Outcome Measures Data:
  Muscle strength values recorded using the hand-held dynamometer for each muscle group (shoulder flexors, abductors, internal rotators, external rotators).
  Proprioception data measured by the laser pointer-assisted joint position reproduction test, including the distance (in millimeters) between the initial and reproduced positions for both shoulder flexion and abduction.
  Group Assignment Data:
  Whether the participant was assigned to the mobilization group or the sham intervention group.
  Intervention Data:
  Details of the intervention received, including whether they underwent shoulder mobilization or placebo procedure.
  Timing of Measurements:
  Pre- and post-intervention data for both muscle strength and proprioception assessments.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD and supporting information will be made available starting from the date of publication of the study's results. The data will be accessible for 5 years from the publication date to allow for ample time for further analysis, replication studies, or meta-analysis by other researchers.
Access Criteria: Who Can Access:
  * Researchers, academics, and institutional partners with a legitimate research purpose.
  * Regulatory agencies or health organizations.
  What They Can Access:
  * Anonymized IPD (muscle strength, proprioception, demographics).
  * Supporting information (study protocol, SAP,)
  How They Can Access:
  * Data will be shared upon contact with the study team.
  * Interested parties must request access, and data will be provided following review and approval.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a university setting between April and May 2025. All participants provided written informed consent.
Pre-assignment Details: 48 participants were assessed for eligibility and randomized before any intervention was delivered. No dropouts or exclusions occurred.
Groups:
- Mobilization Group: Received passive glenohumeral joint mobilization (inferior, anterior, posterior glides).
- Sham Group: Received simulated mobilization without mechanical input.
Period: Overall Study
Arm/Group | Mobilization Group | Sham Group
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobilization Group | Sham Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Full Range); unit: years] | 21.08 [18 to 24] | 20.91 [18 to 23] | 21 [18 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 24 | 24 | 48
Muscle strength [Median (Inter-Quartile Range); unit: kg]
  Flexion | 17.3 [13.5 to 26.6] | 19.5 [13.1 to 27.3] | 17.6 [13.4 to 27.3]
  Abduction | 17.6 [14.4 to 24.7] | 17.8 [13.4 to 25.6] | 17.6 [14 to 25.2]
  External Rotation | 9.82 [8.27 to 13.1] | 9.4 [8.18 to 14.7] | 9.47 [8.18 to 14.2]
  Internal Rotation | 15.4 [11.3 to 19.5] | 14.6 [9.8 to 19.7] | 14.6 [10.6 to 19.7]
Proprioception Error [Median (Inter-Quartile Range); unit: mm]
  Flexion | 54 [45.3 to 68.3] | 62.8 [48.3 to 80.1] | 57.3 [46.7 to 77]
  Abduction | 86.7 [68.8 to 111] | 85.3 [64.8 to 98.3] | 86.2 [65 to 107]

OUTCOME MEASURES:

1. Primary Outcome: Proprioception
Description: Laser pointer-assisted joint position reproduction test for shoulder:
  A laser pointer is strapped 5 cm above the lateral epicondyle. Participants actively move their arm to a predefined position (90° flexion or abduction), and the laser projection is marked.
  After lowering their arm and closing their eyes, they attempt to replicate the same position.
  The difference between the initial and reproduced positions (in millimeters) is measured
Time Frame: Before the intervention
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Mobilization Group | Sham Group
Number analyzed (Participants) | 24 | 24
mm
  Proprioception Flexion | 54 (20.9) | 62.8 (22.8)
  Proprioception Abduction | 86.7 (32.1) | 85.3 (26.6)

2. Primary Outcome: Proprioception
Description: as for outcome 1
Time Frame: Immediately after intervention
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Mobilization Group | Sham Group
Number analyzed (Participants) | 24 | 24
mm
  Proprioception Flexion | 52.3 (23.9) | 52.2 (78.3)
  Proprioception Abduction | 91.2 (29) | 78.3 (32.5)

3. Secondary Outcome: Muscle Strength
Description: Hand-held dynamometer (Lafayette) Muscle strength will be measured using a hand-held dynamometer (Lafayette). The assessment will focus on the shoulder flexors, abductors, internal rotators, and external rotators. Three measurements for each muscle group will be taken, and the average value will be recorded in kilograms (kg).
Time Frame: Before the intervention
Measure: Median (Standard Deviation); unit: kg
Arm/Group | Mobilization Group | Sham Group
Number analyzed (Participants) | 24 | 24
kg
  Shoulder Flexion | 17.3 (7.59) | 19.5 (9.08)
  Shoulder Abduction | 17.6 (7.32) | 17.8 (7.58)
  Shoulder External Rotation | 9.82 (3.60) | 9.40 (4.10)
  Shoulder Internal Rotation | 15.4 (5.84) | 14.6 (5.91)

4. Secondary Outcome: Muscle Strength
Description: as for outcome 3
Time Frame: Immediately after intervention
Measure: Median (Standard Deviation); unit: kg
Arm/Group | Mobilization Group | Sham Group
Number analyzed (Participants) | 24 | 24
kg
  Shoulder Flexion | 18.3 (8.03) | 18.5 (9.42)
  Shoulder Abduction | 16.6 (6.81) | 16.5 (8.35)
  Shoulder External Rotation | 9.83 (3.05) | 9.95 (4.87)
  Shoulder Internal Rotation | 15.1 (5.86) | 14.2 (6.45)

ADVERSE EVENTS:
Time Frame: Immediately post-intervention (same day)
Description: Participants were monitored during and immediately after the intervention session for adverse events.
Arm/Group | Mobilization Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT06910332/Prot_SAP_000.pdf